CLINICAL TRIAL: NCT06268522
Title: Adjunctive Mindfulness During Opioid Tapering for Patients With Chronic Pain
Brief Title: Adjunctive Mindfulness During Opioid Tapering for patientS With Chronic Pain (The AMOS Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Asimina Lazaridou, PhD, Instructor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023P001582
Record Dates: First submitted 2024-02-02; First posted 2024-02-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Behavioral
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Oriented Recovery Enhancement: (MORE) group (Experimental)
  Interventions: Behavioral: Mindfulness-Oriented Recovery Enhancement: (MORE) group
- Psychoeducation (Placebo Comparator)
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Mindfulness-Oriented Recovery Enhancement: (MORE) group — Mindfulness-Oriented Recovery Enhancement (MORE) is a novel social work intervention and mental training program that unites complementary aspects of mindfulness training.
  Arms: Mindfulness-Oriented Recovery Enhancement: (MORE) group
Behavioral: Psychoeducation — Education on the neurobiology of pain, healthy eating, diet, sleep and stress
  Arms: Psychoeducation

SUMMARY:
This study is a Randomized Controlled Trial exploring the effects of a Mindfulness interventions in reducing pain interference and opioid dose in patients with Chronic Low Back Pain. A total of 200 opioid-using patients with chronic pain, male and female participants will be enrolled, with a need for 160 completers. Patient will be randomly assigned into the Mindfulness-Oriented Recovery Enhancement or the Psychoeducation comparison control group.

ELIGIBILITY:
Inclusion criteria:

* age>18yo
* Chronic Low Back Pain as seen on medical history as well as score of >3 on pain visual analog scale (VAS) at the start of experimental sessions.
* receiving prescription opioids for three or more months and planning to start tapering their opioids with their provider.
* willing to be randomized to one of the two behavioral treatment. Patients referred or self-referred to the study from an outside clinic will also be able to participate (we will be in contact with their prescribing provider)
* able and willing to perform/tolerate pain procedures (e.g., QST)
* able to communicate fluently in English
* able to use a smartphone or laptop for the virtual therapy program

Exclusion criteria:

* Current illicit substance use (e.g marijuana use will be exempted) at screening or during trial as verified by urine toxicology screen and/or self-report for all participants;
* Medical condition known to influence QST or participation in the MORE intervention; serious psychiatric condition;
* regular meditation practice
* cognitive impairment
* pregnancy
* lack of English fluency
* severe OUD
* inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-28 (Actual); Study Completion 2025-06-28 (Actual)

PRIMARY OUTCOMES:
Pain Interference | Baseline, 8 weeks, 3 month and 6 month follow up
  assessed by the Brief pain interventory
Opioid Dose | Baseline, 8 weeks, 3 month and 6 month follow up
  assessed through their medical record

SECONDARY OUTCOMES:
Pain Intensity | Baseline, 8 weeks, 3 month and 6 month follow up
  assessed through the Brief Pain Inventory
Opioid Misuse | Baseline, 8 weeks, 3 month and 6 month follow up
  assessed by the Current Opioid Misuse Measure (COMM)
Opioid Withdrawal | Baseline, 8 weeks, 3 month and 6 month follow up
  assessed by the Opioid Withdrawal Scale (SOWS)
Opioid Craving | Baseline,8 weeks, 3 month and 6 month follow up
  assessed by the single item Opioid Craving

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet the IPD sharing plan